CLINICAL TRIAL: NCT04270110
Title: Assessment of Bone Mineral Density in Patients With Subclinical Hypothyroidism
Acronym: ABMDPSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, kareem mohammed mohammed, resident doctor, Assiut University
Other Study IDs: assessmentofbonemineral
Record Dates: First submitted 2020-01-16; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Subclinical hypothyroïdism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with subclinical hypothyroidism
- Control: Patients with Normal thyroid function

SUMMARY:
This study aims to recognize the effects of subclinical hypothyroidism on bone mineral density, Not many studies were done on this subject

DETAILED DESCRIPTION:
A lot of different factors are necessary for the harmonious development as well as normal functioning of skeleton: genetic conditions, hormonal and metabolic homeostasis, balanced diet, mechanical load. Any disturbances of those agents can lead to serious and dangerous consequences like length reduction, deformations, and fractures. Their results depend, between other, on one's age, type of disorder and its duration.

* There are a lot of endocrinological reasons of secondary osteoporosis (for example: Cushing's syndrome, hyperparathyroidism, hypogonadism, acromegaly, diabetes mellitus, hypothyroidism etc..

Any changes of normal thyroid function and Thyroid stimulating hormones (TSH) directly affects the remodeling of bone through TSH receptor found on osteoblast and osteoclast precursor cells.

TSH has a positive correlation with body mass index (BMI) in women; though, this correlation is insignificant in male. Women having subclinical hypothyroidism have reduced femoral neck bone mineral density (BMD). The variations in thyroid function are primary, while changes in body weight and bones are secondary. The physiological variation of thyroid hormones is associated with changes in BMD and non vertebral fracture risk in healthy postmenopausal women.

The definition of osteoporosis by the world health organization (WHO) is densitometric and non-clinical and is based on the measurement of bone mass and dexa method in the spine or hip. There is still controversy about the relation between thyroid hormones, osteoporosis and BMD in female hypothyroid patients. This study aims to fill the gaps in our understanding of impact of subclinical hypothyroid disorder on bone densitometry.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients with subclinical hypothyroidism with the level of TSH values above 4.0 mU/l.and normal values of thyroxine (T4) and triiodothyronine (T3).

Exclusion Criteria:

* Diabetes mellitus
* Cushing
* hyperparathrodisim
* CKD .patients on corticosteroid therapy.
* Inflammatory conditions as rheumatoid arthritis,Systemic Lupus, Crohn's disease, ulcerative colitis
* Haematological conditions as multiple myeloma, Myeloproliferative disorders
* Vitamin D deficiency
* Males aged more than 55 years old
* Postmenopausal females will also be excluded in this study

Max Age: 55 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients: -case: patients with subclinical hypothyroidism.
  * control: patients with normal thyroid function
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
association between thyroid function parameters and bone densitometry | 1 year
  association of Subclinical hypothyroidism which represents a state with increased values of thyroid stimulating hormone (TSH) and normal values of thyroxine (T4) and triiodothyronine (T3). The disorder is asymptomatic, and the diagnosis is made based on the results of laboratory findings when the level of TSH reaches values above 4.0 mU/ with osteoporesis disorder on bone densitometry. Dual x-ray absorptiometry (DXA) is currently the standard for assessing bone mineral density (BMD), in this study dxa scan will be used on the forearm to assess T score and Z score.

SECONDARY OUTCOMES:
- To detect early stages of bone affection in patients with subclinical hypothyroidism | 1 year
  - To detect early stages of bone affection in patients with subclinical hypothyroidism

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakatos P. Thyroid hormones: beneficial or deleterious for bone? Calcif Tissue Int. 2003 Sep;73(3):205-9. doi: 10.1007/s00223-002-0027-8. PMID 14667131
- See also: Thyroid Hormones: Beneficial or Deleterious for Bone? — https://link.springer.com/article/10.1007/s00223-002-0027-8